CLINICAL TRIAL: NCT05202262
Title: A Randomized, Double-Blind, Parallel Group, Multicenter 24 Week Study to Assess the Efficacy and Safety of Budesonide and Formoterol Fumarate Metered Dose Inhaler Relative to Budesonide Metered Dose Inhaler and Open-Label Symbicort® Turbuhaler® in Participants With Inadequately Controlled Asthma (VATHOS).
Brief Title: A 24-Week Efficacy and Safety Study to Assess Budesonide and Formoterol Fumarate Metered Dose Inhaler in Adult and Adolescent Participants With Inadequately Controlled Asthma (VATHOS)
Acronym: VATHOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5982C00006; 2024-513568-24-00 (Registry Identifier: CTIS); 2021-002026-24 (EudraCT Number)
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Open Label for Symbicort TBH
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BFF MDI 320/9.6 μg (Experimental): Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), 320/9.6 μg
  Interventions: Drug: BFF MDI 320/9.6 μg
- BFF MDI 160/9.6 μg (Experimental): Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), 160/9.6 μg
  Interventions: Drug: BFF MDI 160/9.6 μg
- BD MDI 320 μg (Experimental): Budesonide MDI (BD MDI), 320 μg
  Interventions: Drug: BD MDI 320 μg
- Open-label Symbicort TBH 320/9 μg (Active Comparator): Open-Label Comparator Symbicort Turbuhaler 320/9 μg
  Interventions: Drug: Open-label Symbicort TBH 320/9 μg

INTERVENTIONS:
Drug: BFF MDI 320/9.6 μg — Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), 320/9.6 μg
  Other Names: BFF
  Arms: BFF MDI 320/9.6 μg
Drug: BFF MDI 160/9.6 μg — Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), 160/9.6 μg
  Other Names: BFF
  Arms: BFF MDI 160/9.6 μg
Drug: BD MDI 320 μg — Budesonide MDI (BD MDI), 320 μg
  Other Names: BD
  Arms: BD MDI 320 μg
Drug: Open-label Symbicort TBH 320/9 μg — Open-label Symbicort Turbuhaler 320/9 μg
  Other Names: Symbicort TBH
  Arms: Open-label Symbicort TBH 320/9 μg

SUMMARY:
This is a 24 week study to evaluate the efficacy and safety of budesonide and formoterol fumarate metered dose inhaler in adults and adolescents with inadequately controlled asthma.

DETAILED DESCRIPTION:
This is a Phase III randomized, double-blind, active comparison, parallel group, multicenter study comparing BFF MDI 320/9.6 μg to BD MDI 320 µg and open-label Symbicort TBH 320/9 μg in adult and adolescent participants who have asthma which remains inadequately controlled (ACQ-7 total score ≥ 1.5) despite treatment with medium dose ICS or ICS/LABA. Budesonide and Formoterol Fumarate MDI 160/9.6 μg is included in this study to evaluate dose response by comparing to BFF MDI 320/9.6 μg. All doses represent the sum of 2 actuations. All study interventions will be administered BID for 24 weeks.

This study will be conducted at approximately 125 sites worldwide and will randomize approximately 630 adult and adolescent participants.

ELIGIBILITY:
Inclusion Criteria:

1. 12 to 80 years of age, male and female, BMI <40 kg/m2; females must be not of childbearing potential or using a form of highly effective birth control.
2. Participants who have a documented history of physician-diagnosed asthma ≥ 6 months prior to Visit 1, according to GINA guidelines [GINA 2020]. Healthcare records for one year prior to Visit 1 must be provided for adolescent participants (12 to < 18 years of age) to ensure consistent evaluation and follow-up of treatment in those participants.
3. Participants who have been regularly using a stable daily ICS or an ICS/LABA regimen (including a stable ICS dose), with the ICS doses, for at least 8 weeks prior to Visit 1.
4. ACQ-7 total score ≥ 1.5 at Visits 1 and 4.
5. Pre-bronchodilator/pre-dose FEV1 <90% predicted normal value at Visits 1, 2 and 3, and a pre-dose FEV1 of 50% to 90% at Visit 4 (pre-randomization).
6. Reversibility to albuterol, defined as a post-albuterol increase in FEV1 of ≥ 12% and ≥ 200 mL for participants ≥ 18 years of age OR a post-albuterol increase in FEV1 of ≥ 12% for participants 12 to < 18 years of age, either in the 12 months prior to Visit 1 or at Visit 2 or Visit 3.
7. A pre-bronchodilator/pre-dose FEV1 at Visits 2, 3, and 4 that have not changed 20% or more (increase or decrease) from the pre-bronchodilator/pre-dose FEV1 recorded at the previous visit.
8. Asthma stability during run-in based on Investigator discretion using the symptom worsening assessment.
9. Willing and, in the opinion of the Investigator, able to adjust current asthma therapy, as required by the protocol.
10. Demonstrate acceptable MDI administration technique.
11. eDiary compliance ≥ 70% during screening, defined as completing the daily eDiary and answering "Yes" to taking 2 puffs of run-in BD MDI for any 10 mornings and 10 evenings in the last 14 days prior to randomization.

Exclusion Criteria:

1. Life-threatening asthma as defined as a history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma related syncopal episode(s).
2. Any respiratory infection or asthma exacerbation treated with systemic corticosteroids and/or additional ICS treatment in the 8 weeks prior to Visit 1 and throughout the Screening Period.
3. Hospitalization for asthma within 8 weeks of Visit 1.
4. Historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular, hepatic, renal, hematological, neurological, endocrine, gastrointestinal, or pulmonary (eg, active tuberculosis, bronchiectasis, pulmonary eosinophilic syndromes, and COPD). Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the participant at risk through participation, or that could affect the efficacy or safety analysis.
5. Known history of drug or alcohol abuse within 12 months of Visit 1.
6. Unresectable cancer that has not been in complete remission for at least 5 years prior to Visit 1.
7. Participation in another clinical study with a study intervention administered in the last 30 days or 5 half-lives, whichever is longer. Any other study intervention that is not identified in this protocol is prohibited for use during study duration.
8. Previous or current randomization into studies within the AEROSPHERE program including KALOS, LOGOS, VATHOS, LITHOS, or any glycopyrronium studies (PT001).
9. Use of a nebulizer or a home nebulizer for receiving asthma medications.
10. Do not meet the stable dosing period prior to Visit 1 or unable to abstain from protocol-defined prohibited medications during Screening and Treatment Periods.
11. Receipt of COVID-19 vaccine (regardless of vaccine delivery platform, eg, vector, lipid nanoparticle) < 7 days prior to Visit 1 (from last vaccination or booster dose).
12. Participants with known hypersensitivity to beta2-agonists, corticosteroids, or any component of the MDI.
13. Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, vital signs, or ECG, which in the opinion of the Investigator, may put the participant at risk because of his/her participation in the study.
14. Current smokers, former smokers with > 10 pack-years history, or former smokers who stopped smoking < 6 months prior to Visit 1 (including all forms of tobacco, e-cigarettes or other vaping devices, and marijuana).
15. Planned hospitalization during the study.
16. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
17. Study Investigators, sub-Investigators, coordinators, and their employees or immediate family members.
18. Judgment by the Investigator that the participant is unlikely to comply with study procedures, restrictions, and requirements.
19. For women only - currently pregnant (confirmed with positive highly sensitive urine pregnancy test), breast-feeding, or planned pregnancy during the study or not using acceptable contraception measures, as judged by the Investigator.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (115):
- United States (59):
  - Research Site, Chandler, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Fresno, California
  - Research Site, Huntington Beach, California
  - Research Site, La Palma, California
  - Research Site, Lincoln, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Denver, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Cutler Bay, Florida
  - Research Site, DeLand, Florida
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Peoria, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, White Marsh, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Columbia, Missouri
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Kalispell, Montana
  - Research Site, Missoula, Montana
  - Research Site, Bellevue, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, North Las Vegas, Nevada
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Skillman, New Jersey
  - Research Site, Gastonia, North Carolina
  - Research Site, Monroe, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Forney, Texas
  - Research Site, Houston, Texas
  - Research Site, Red Oak, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Victoria, Texas
  - Research Site, Waco, Texas
  - Research Site, Williamsburg, Virginia
  - Research Site, Milwaukee, Wisconsin
- Canada (12):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Kamloops, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Stouffville, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Germany (9):
  - Research Site, Berlin
  - Research Site, Frankfurt am Main
  - Research Site, Landsberg
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, München-Pasing
  - Research Site, Schleswig
  - Research Site, Wiesbaden
  - Research Site, Witten
- Italy (6):
  - Research Site, Brescia
  - Research Site, Mantova
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Rome
  - Research Site, Tradate
- Japan (20):
  - Research Site, Chūōku
  - Research Site, Fukui-shi
  - Research Site, Fukuoka
  - Research Site, Himeji-shi
  - Research Site, Kagoshima
  - Research Site, Kishiwada-shi
  - Research Site, Kodaira-shi
  - Research Site, Kokubunji-shi
  - Research Site, Kusatsu-shi
  - Research Site, Kyoto
  - Research Site, Mizunami-shi
  - Research Site, Obihiro-shi
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Setagaya-ku
  - Research Site, Shibuya-ku
  - Research Site, Toon-shi
  - Research Site, Toshima-ku
  - Research Site, Utsunomiya
  - Research Site, Yokohama
- Spain (7):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Santiago de Compostela
  - Research Site, Vigo
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5982C00006&attachmentIdentifier=cea6c9d8-e6e7-4bb9-b601-c8925bd2cf01&fileName=D5982C00006_VATHOS_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who have asthma which remains inadequately controlled (ACQ-7 total score ≥ 1.5) despite treatment with medium dose ICS or ICS/LABA were recruited at 147 sites across 7 countries. Participants were randomized in a 1:2:2:2 scheme to BFF MDI 160/9.6 μg, BFF MDI 320/9.6 μg, BD MDI 320 μg, or open-label Symbicort. Randomization was stratified by baseline asthma treatment and age. The treatment period was 24 weeks in duration with up to 8 in-clinic visits during screening and treatment.
Pre-assignment Details: All participants were on stable daily medium dose ICS or ICS/LABA for at least 8 weeks prior to Visit 1. After meeting the screening eligibility criteria, participants discontinued medium dose ICS or ICS/LABA at Visit 1 and initiated run-in BD MDI 320 µg taking BID until the randomization visit. A total of 581 patients were treated and included in the safety population. Of the 645 initially randomized, 64 were excluded (60 from 11 sites with GCP violation and 4 who did not receive therapy).
Groups:
- BFF MDI 160/9.6 g: Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), 160/9.6 μg
- BFF MDI 320/9.6 g: Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), 320/9.6 μg
- BD MDI 320 g: Budesonide MDI (BD MDI), 320 μg
- Symbicort TBH 320/9 g: Open-Label Comparator Symbicort Turbuhaler 320/9 μg
Period: Overall Study
Arm/Group | BFF MDI 160/9.6 g | BFF MDI 320/9.6 g | BD MDI 320 g | Symbicort TBH 320/9 g
Started | 88 | 163 | 168 | 162
Completed | 81 | 150 | 155 | 151
Not Completed | 7 | 13 | 13 | 11
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 4 | 0
Not completed — Physician Decision | 3 | 3 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Development of withdrawal Criteria | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 5 | 4
Not completed — Various Reasons | 2 | 5 | 3 | 4
Not completed — Failure to meet randomization criteria | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Efficacy Set is defined as all participants who are randomized to study intervention and receive any amount of randomized study intervention. It excludes 6 participants who were randomized before or concurrently in another study.
Groups:
- Total: Total of all reporting groups
Arm/Group | BFF MDI 160/9.6 g | BFF MDI 320/9.6 g | BD MDI 320 g | Symbicort TBH 320/9 g | Total
Number analyzed (Participants) | 87 | 162 | 166 | 160 | 575
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (17.2) | 49.7 (15.8) | 49.0 (15.2) | 51.3 (15.3) | 49.9 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 101 | 108 | 101 | 358
  Male | 39 | 61 | 58 | 59 | 217
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 9 | 16 | 17 | 24 | 66
  Asian | 9 | 22 | 18 | 19 | 68
  White | 64 | 119 | 122 | 112 | 417
  Other | 5 | 5 | 9 | 5 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  Global: Canada | 6 | 13 | 10 | 8 | 37
  Global: Germany | 27 | 33 | 39 | 30 | 129
  Global: Italy | 4 | 4 | 1 | 6 | 15
  Global: Japan | 4 | 12 | 8 | 9 | 33
  Global: Spain | 3 | 6 | 7 | 6 | 22
  Global: United States | 40 | 88 | 97 | 92 | 317
  Global: Vietnam | 3 | 6 | 4 | 9 | 22
Prior asthma medication [Count of Participants; unit: Participants]
  ICS | 11 | 17 | 20 | 19 | 67
  ICS/LABA | 76 | 145 | 145 | 141 | 507
  ICS/LAMA/LABA | 0 | 0 | 1 | 0 | 1
Baseline reversibility (%) [Mean (Standard Deviation); unit: Percentage] — Baseline reversibility (%): ((Post-Albuterol FEV1 - Pre-Albuterol FEV1)/ Pre-Albuterol FEV1) x 100
  Percentage | 18.5 (11.3) | 17.5 (12.8) | 19.9 (11.0) | 20.0 (15.9) | 19.0 (13.1)
Baseline pre-bronchodilator FEV1 (L) [Mean (Standard Deviation); unit: Liter] — Baseline pre-bronchodilator FEV1 (L) is the mean of the pre-dose FEV1 at -60 and -30 minutes on Day 1, using the best effort at each timepoint. Population: Two participants have missing pre-bronchodilator FEV1 at baseline.
  Liter
    number analyzed (Participants) | 87 | 161 | 166 | 159 | 573
    (all) | 2.315 (0.666) | 2.163 (0.666) | 2.132 (0.561) | 2.103 (0.589) | 2.160 (0.618)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve 0 to 3 Hours (AUC0-3) at Week 24
Description: Change from baseline in forced expiratory volume in 1 second (FEV1) area under the curve 0 to 3 hours (AUC0-3) at Week 24. FEV1 AUC0-3 is calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time to report the result in liters. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: At Week 24
Population: The Efficacy Set is defined as all participants who are randomized to study intervention and receive any amount of randomized study intervention. Participants are analyzed according to the treatment assigned at randomization, regardless of the actual treatment received. Only subjects with non-missing baseline covariates used in the analysis model are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liter
Groups:
- Symbicort TBH 320/9 μg: Open-Label Comparator Symbicort Turbuhaler 320/9 μg
Arm/Group | BFF MDI 160/9.6 μg | BFF MDI 320/9.6 μg | BD MDI 320 μg | Symbicort TBH 320/9 μg
Number analyzed (Participants) | 83 | 155 | 160 | 155
Liter | 0.276 (0.0300) | 0.240 (0.0219) | 0.067 (0.0216) | 0.240 (0.0220)
Statistical Analysis 1: Comparison: BFF MDI 320/9.6 μg vs BD MDI 320 μg; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.173, 95% CI 2-sided [0.112 to 0.233], Standard Error of Mean 0.0308 — An increase in estimate favors study drug. The model includes treatment, visit, prior maintenance medication, treatment-by-visit interaction, baseline trough FEV1, and percent Albuterol reversibility

2. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 at Week 24
Description: Change from baseline in morning pre-dose trough FEV1 at Week 24. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: At 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | BFF MDI 160/9.6 μg | BFF MDI 320/9.6 μg | BD MDI 320 μg | Symbicort TBH 320/9 μg
Number analyzed (Participants) | 84 | 155 | 161 | 155
Liter | 0.125 (0.0293) | 0.099 (0.0215) | 0.038 (0.0211) | 0.131 (0.0216)
Statistical Analysis 1: Comparison: BFF MDI 320/9.6 μg vs BD MDI 320 μg; Test type: Superiority; p = 0.0447, ANCOVA; Mean Difference (Final Values) = 0.061, 95% CI 2-sided [0.001 to 0.120], Standard Error of Mean 0.0302 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Onset of Action on Day 1: Absolute Change in FEV1 at 5 Minutes on Day 1
Description: Onset of action on Day 1: Absolute change in FEV1 at 5 minutes on Day 1. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: On Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | BFF MDI 160/9.6 μg | BFF MDI 320/9.6 μg | BD MDI 320 μg | Symbicort TBH 320/9 μg
Number analyzed (Participants) | 84 | 159 | 158 | 156
Liter | 0.236 (0.0167) | 0.184 (0.0122) | 0.041 (0.0121) | 0.161 (0.0123)
Statistical Analysis 1: Comparison: BFF MDI 320/9.6 μg vs BD MDI 320 μg; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.144, 95% CI 2-sided [0.110 to 0.177], Standard Error of Mean 0.0172 — An increase in estimate favors study drug. The model includes treatment, timepoint, prior maintenance medication, treatment-by-timepoints interaction, baseline tFEV1, and % Albuterol reversibility

4. Secondary Outcome: Change From Baseline in the Mean Number of Puffs of Rescue Medication Use (Puffs/Day) Over 24 Weeks
Description: Change from baseline in the mean number of puffs of rescue medication use (puffs/day) over 24 Weeks. Baseline is the average during the last 7 days before randomization. Over 24 weeks is the average from randomization up to week 24. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: Over 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs/Day
Arm/Group | BFF MDI 160/9.6 μg | BFF MDI 320/9.6 μg | BD MDI 320 μg | Symbicort TBH 320/9 μg
Number analyzed (Participants) | 85 | 157 | 163 | 153
Puffs/Day | -0.350 (0.1061) | -0.481 (0.0781) | -0.213 (0.0764) | -0.443 (0.0791)
Statistical Analysis 1: Comparison: BFF MDI 320/9.6 μg vs BD MDI 320 μg; Test type: Superiority; p = 0.0146, ANCOVA; Mean Difference (Final Values) = -0.268, 95% CI 2-sided [-0.482 to -0.053], Standard Error of Mean 0.1092 — A decrease in estimate favors study drug. The model includes treatment, 4-week interval, their interaction, prior maintenance medication, severe asthma exacerbation history, baseline daily rescue use, baseline tFEV1, and % Albuterol reversibility

5. Secondary Outcome: Percentage of Responders in ACQ-7 (≥ 0.5 Decrease Equals Response) at Week 24
Description: Percentage of responders in ACQ-7 at Week 24, where responders are defined as participants with a ≥0.5 decrease in total score from baseline. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BFF MDI 160/9.6 μg | BFF MDI 320/9.6 μg | BD MDI 320 μg | Symbicort TBH 320/9 μg
Number analyzed (Participants) | 82 | 155 | 161 | 154
Percentage of participants | 70.7 | 68.4 | 62.7 | 71.4
Statistical Analysis 1: Comparison: BFF MDI 320/9.6 μg vs BD MDI 320 μg; Test type: Superiority; p = 0.2977, Regression, Logistic; Odds Ratio (OR) = 1.283, 95% CI 2-sided [0.803 to 2.052] — An odds ratio greater than 1 favors study drug. The model includes treatment, prior maintenance medication, baseline instrument score, baseline tFEV1, and % Albuterol reversibility

6. Secondary Outcome: Percentage of Responders in ACQ-5 (≥ 0.5 Decrease Equals Response) at Week 24
Description: Percentage of responders in ACQ-5 at Week 24, where responders are defined as participants with a ≥0.5 decrease in total score from baseline. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BFF MDI 160/9.6 μg | BFF MDI 320/9.6 μg | BD MDI 320 μg | Symbicort TBH 320/9 μg
Number analyzed (Participants) | 82 | 155 | 161 | 154
Percentage of participants | 75.6 | 71.6 | 65.8 | 68.8
Statistical Analysis 1: Comparison: BFF MDI 320/9.6 μg vs BD MDI 320 μg; Test type: Superiority; p = 0.2477, Regression, Logistic; Odds Ratio (OR) = 1.332, 95% CI 2-sided [0.819 to 2.166] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Percentage of Responders in the Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ(s)+12) (≥ 0.5 Increase Equals Response) at Week 24
Description: Percentage of responders in the Asthma Quality of Life Questionnaire for 12 years and older (AQLQ(s)+12) at Week 24, where responders are defined as participants with a ≥0.5 increase in total score from baseline. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BFF MDI 160/9.6 μg | BFF MDI 320/9.6 μg | BD MDI 320 μg | Symbicort TBH 320/9 μg
Number analyzed (Participants) | 79 | 149 | 157 | 147
Percentage of participants | 53.2 | 57.7 | 47.1 | 50.3
Statistical Analysis 1: Comparison: BFF MDI 320/9.6 μg vs BD MDI 320 μg; Test type: Superiority; p = 0.0194, Regression, Logistic; Odds Ratio (OR) = 1.770, 95% CI 2-sided [1.097 to 2.858] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Rate of Severe Asthma Exacerbation (Pooled LITHOS and VATHOS Data) During the Treatment Period (up to 24 Weeks)
Description: As requested by a Health Authority, data from VATHOS and LITHOS (NCT05755906), two studies originally designed to assess lung function, were pooled to analyze the annualized rate of severe asthma exacerbations. This analysis was prespecified, uses data up to 12 weeks for LITHOS and 24 weeks for VATHOS, and was incorporated into the multiple testing procedure. An exacerbation is considered severe if it results in at least one of the following: a course of systemic corticosteroids (SCS) for ≥3 consecutive days to treat symptoms of asthma worsening, an ER or urgent care visit due to asthma requiring treatment with SCS, an in-patient hospitalization due to asthma, or death related to asthma. Treatment policy is implemented to handle all intercurrent events except for initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is used.
Time Frame: 24 Weeks
Population: The Efficacy Set is defined as all participants in VATHOS and LITHOS (NCT05755906) who are randomized to study intervention and receive any amount of randomized study intervention. Participants are analyzed according to the treatment assigned at randomization, regardless of the actual treatment received. Only subjects with non-missing baseline covariates used in the analysis model are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Exacerbations/year
Groups:
- BFF MDI 160/9.6 μg or 320/9.6 μg: Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), 160/9.6 μg BID (320/19.2μg/day) or Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), 320/9.6 μg BID (640/19.2μg/day)
- BD MDI 160 μg or 320 μg: Budesonide (BD) metered-dose inhaler (MDI), 160 μg BID (320 μg/day) or Budesonide (BD) metered-dose inhaler (MDI), 320 μg BID (640 μg/day)
Arm/Group | BFF MDI 160/9.6 μg or 320/9.6 μg | BD MDI 160 μg or 320 μg
Number analyzed (Participants) | 425 | 335
Exacerbations/year | 0.35 (0.05) | 0.42 (0.07)
Statistical Analysis 1: Comparison: BFF MDI 160/9.6 μg or 320/9.6 μg vs BD MDI 160 μg or 320 μg; Test type: Superiority; p = 0.3610, Regression, Negative Binomial; Rate Ratio = 0.82, 95% CI [0.54 to 1.25] — A rate ratio below 1 favors study drug. The model includes budesonide dose, formoterol dose, study, severe asthma exacerbation history, prior maintenance medications, baseline tFEV1, % Albuterol reversibility, and region

9. Secondary Outcome: Rate of Severe Asthma Exacerbation During the Treatment Period (up to 24 Weeks)
Description: Annualized rate of severe asthma exacerbation during the treatment period (up to 24 Weeks). An asthma exacerbation will be considered severe if it results in at least one of the following: a course of systemic corticosteroids for at least 3 consecutive days to treat symptoms of asthma worsening, an ER or urgent care visit due to asthma that required treatment with systemic corticosteroids, an in-patient hospitalization due to asthma, or death related to asthma.
  Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Exacerbations/year
Arm/Group | BFF MDI 160/9.6 μg | BFF MDI 320/9.6 μg | BD MDI 320 μg | Symbicort TBH 320/9 μg
Number analyzed (Participants) | 87 | 161 | 166 | 159
Exacerbations/year | 0.26 (0.08) | 0.36 (0.07) | 0.35 (0.07) | 0.41 (0.07)
Statistical Analysis 1: Comparison: BFF MDI 320/9.6 μg vs BD MDI 320 μg; Test type: Superiority; p = 0.9473, Regression, Negative Binomial; Rate Ratio = 1.02, 95% CI 2-sided [0.61 to 1.70] — A rate ratio lower than 1 favors study drug. The model includes treatment, severe asthma exacerbation history, prior maintenance medications, baseline tFEV1, % Albuterol reversibility, and region

ADVERSE EVENTS:
Time Frame: From the date of first dose of IP up to and including 1 day following the date of last IP dose, up to 24 weeks.
Description: Adverse events were reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative). The Investigator and any designees were responsible for detecting, documenting, and recording events that meet the definition of an AE.
  The Safety Set is defined as the Efficacy Set, but it also includes the 6 participants who were randomized multiple times at sites or studies
Arm/Group | BFF MDI 160/9.6 g | BFF MDI 320/9.6 g | BD MDI 320 g | Symbicort TBH 320/9 g
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/163 | 0/168 | 0/162
Serious Adverse Events (participants affected / at risk) | 3/88 | 3/163 | 1/168 | 7/162
Other Adverse Events (participants affected / at risk) | 31/88 | 45/163 | 40/168 | 39/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BFF MDI 160/9.6 g (N=88) | BFF MDI 320/9.6 g (N=163) | BD MDI 320 g (N=168) | Symbicort TBH 320/9 g (N=162)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BFF MDI 160/9.6 g (N=88) | BFF MDI 320/9.6 g (N=163) | BD MDI 320 g (N=168) | Symbicort TBH 320/9 g (N=162)
Bronchitis bacterial (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Covid-19 (Infections and infestations) | 3 (3) | 15 (15) | 8 (8) | 11 (11)
Nasopharyngitis (Infections and infestations) | 12 (13) | 15 (17) | 15 (20) | 13 (19)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 8 (12) | 12 (15) | 9 (10)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 5 (5)
Gout (Metabolism and nutrition disorders) | 2 (4) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT05202262/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT05202262/SAP_001.pdf